CLINICAL TRIAL: NCT05155241
Title: A Randomized Controlled Trial Evaluating an Online Intervention Based on the Trans-Theoretical Model in Increasing Seasonal Influenza Vaccination Among Community Dwelling People Aged ≥65 Years
Brief Title: A Randomized Controlled Trial Evaluating an Online Intervention in Increasing Seasonal Influenza Vaccination Among Community Dwelling People Aged ≥65 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17180411
Record Dates: First submitted 2021-12-01; First posted 2021-12-13 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Vaccination Refusal
MeSH Terms: conditions — Vaccination Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will watch an online health promotion video tailored to their current stage of change related to SIV uptake once every two weeks for four times (at week 0, 2, 4, and 6)
  Interventions: Behavioral: online health promotion video
- Control (Active Comparator): Participants will watch a same online video providing general advices related to SIV at week 0, 2, 4, and 6
  Interventions: Behavioral: Control (same online health promotion video)

INTERVENTIONS:
Behavioral: online health promotion video — Participants will watch an online health promotion video tailored to their current stage of change related to seasonal influenza vaccination uptake once every two weeks for four times (at week 0, 2, 4, and 6)
  Arms: Intervention
Behavioral: Control (same online health promotion video) — Participants will watch a same online video providing general advices related to seasonal influenza vaccination at week 0, 2, 4, and 6
  Arms: Control

SUMMARY:
A non-blinded two-arm parallel randomized controlled trial will be conducted. Inclusion criteria are: 1) aged ≥65 years, 2) having Hong Kong ID, 3) Chinese speaking, 4) willing to be followed up by telephone, 5) having a smartphone, and 6) have not received SIV for the incoming flu season. Exclusion criteria include: 1) cognitive impairment, blindness or deafness, 2) not able to communicate with others effectively, and 3) with known contradictions of SIV (allergic to previous SIV, diagnosed/suspected egg allergy, with bleeding disorder or on warfarin). A total of 396 participants will be randomly assigned to either the intervention group (n=198) or the control group (n=198). Intervention group will watch an online health promotion video tailored to their current stage of change related to SIV uptake once every two weeks for four times (at week 0, 2, 4, and 6).

Participants in the control group will watch a same online video providing general advices related to SIV at week 0, 2, 4, and 6. All participants will be followed up by telephone 3 and 6 months after the baseline survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years,
* Having Hong Kong ID
* Chinese speaking
* Willing to be followed up by telephone
* Having a smartphone
* Have not received seasonal influenza vaccination for the incoming flu season

Exclusion Criteria:

* Cognitive impairment, blindness or deafness,
* Not able to communicate with others effectively
* With known contradictions of seasonal influenza vaccination listed by the Centre for Health Protection (allergic to previous SIV, diagnosed/suspected egg allergy, with bleeding disorder or on warfarin)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 396 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Seasonal influenza vaccination uptake | 6 months
  Self-reported uptake of one dose of seasonal influenza vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Wang Z, Chan PS, Fang Y, Yu FY, Ye D, Zhang Q, Wong MCS, Mo PKH. Chatbot-Delivered Online Intervention to Promote Seasonal Influenza Vaccination During the COVID-19 Pandemic: A Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2332568. doi: 10.1001/jamanetworkopen.2023.32568. PMID 37695585